CLINICAL TRIAL: NCT03140943
Title: Single Arm, Multicentre Study of Carfilzomib in Combination With Thalidomide and Dexamethasone (CaTD) in Patients With Relapsed and/or Refractory Multiple Myeloma (RRMM)
Brief Title: Carfilzomib Thalidomide and Dexamethasone in Patients With Relapsed and/or Refractory Multiple Myeloma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Collaborators: The Australasian Leukaemia & Lymphoma Group (ALLG) (Unknown); International Myeloma Foundation (Other); Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMN002
Record Dates: First submitted 2017-04-13; First posted 2017-05-04 (Actual); Last update posted 2017-11-06 (Actual); Status verified 2017-02

CONDITIONS: Relapsed and/or Refractory Multiple Myeloma
Keywords: carfilzomib
MeSH Terms: interventions — carfilzomib; Thalidomide; Dexamethasone

STUDY DESIGN:
Intervention Model Description: All patients will continue treatment for 18 cycles (12 induction cycles, 6 maintenance cycles) unless development of adverse events that require early cessation of treatment. Patients will be followed up for progression and survival until 1 year following the completion of the last patient's final cycle of induction therapy.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Carfilzomib, Thalidomide and Dexamethasone (Experimental)
  Interventions: Drug: Carfilzomib, Thalidomide and Dexamethasone

INTERVENTIONS:
Drug: Carfilzomib, Thalidomide and Dexamethasone — Carfilzomib will be given on days 1,2,8,9,15,16 in a 4-week (28 day) cycle during induction cycles 1-12, followed by days 1,2,15,16 in a 4-week cycle during maintenance cycles 13-18 (section 4.0) Dexamethasone, 40mg po will be given on days 1,8,15, 22 in a 4-week cycle during induction cycles 1-12, followed by days 1,15, in a 4-week cycle during maintenance cycles 13-18.
  Thalidomide, 100mg po will be given daily during induction cycles 1-12 only.

SUMMARY:
All patients with multiple myeloma (MM) are destined to relapse even with the best available approved agents. Median OS from diagnosis in the current era is reported at 5.4 years. Given that myeloma remains an incurable disease, future improved OS is therefore reliant on the expansion of salvage options for patients with RRMM.

Carfilzomib (formerly PR-171) is a tetrapeptide epoxyketone-based irreversible inhibitor of the 20S proteasome. This second-generation proteasome inhibitor (PI) is structurally and mechanistically different to the dipeptide boronic acid PI, bortezomib. Compared to bortezomib, carfilzomib showed less off-target activity that may account for the reduced myelosuppression and reduced neuropathy that is observed compared to bortezomib. As monotherapy, carfilzomib has demonstrated robust and durable activity in heavily pre-treated patients with RRMM in phase I and II trials The idea of combining a PI and an immunomodulatory drug (IMiD) such as thalidomide or lenalidomide is attractive in MM due to the efficacy previously demonstrated with combination bortezomib, thalidomide and dexamethasone. Such efficacy obviates the need for chemotherapy that is known to induce genetic instability and in turn gives rise to secondary cancers. In combination with lenalidomide (25mg), Niesvizky and colleagues have demonstrated a maximum planned dose (MPD) of carfilzomib as 20/27 mg/m2 with promising safety and efficacy. Combination carfilzomib and thalidomide, as opposed to lenalidomide, is practically a more affordable regimen that will be more applicable to the Asia-Pacific region.

DETAILED DESCRIPTION:
All patients will continue treatment for 18 cycles (12 induction cycles, 6 maintenance cycles) unless development of adverse events that require early cessation of treatment. Patients will be followed up for progression and survival until 1 year following the completion of the last patient's final cycle of induction therapy.

Proteasome inhibitors and IMiDs have different but overlapping mechanisms of anti-MM activity. In the clinical setting, both proteasome inhibitors and IMiDs enhance the activity of dexamethasone, and synergy has previously been demonstrated between the first in class proteasome inhibitor, bortezomib[16] and the immunomodulatory drug lenalidomide[17]. Relative to bortezomib, carfilzomib demonstrated increased apoptosis in MM cell lines, and induce high ORR in both bortezomib-naïve and resistant patients.

We hypothesise that carfilzomib will induce a synergistic anti-myeloma activity when combined with the first in class immunomodulatory drug thalidomide, and dexamethasone. Thalidomide is a cheaper immunomodulatory drug that is more accessible in the Asia-Pacific region compared to lenalidomide. This makes the combination of carfilzomib, thalidomide and dexamethasone a more viable salvage option for patients in this region.

In the PX-171-006 study, combination carfilzomib lenalidomide and dexamethasone induced a CR/VGPR in 59% of patients. The maximum per protocol doses of carfilzomib (27g/m2) was used safely with full dose lenalidomide (25mg po daily days 1-21 every 28 days) and dexamethasone (40 mg po weekly), and the MTD of carfilzomib was not reached.

Carfilzomib 56mg/m2 was tolerable in phase II trials and induced durable responses in patients with relapsed and/or refractory myeloma. The most common grade 3/4 side effects of lymphopenia (43%), thrombocytopenia (32%), hypertension (25%), and pneumonia (18%) are not expected to overlap significantly with the expected side effects of thalidomide [15].

We will combine carfilzomib 20/56mg per m2 in combination with thalidomide 100mg daily and dexamethasone 40mg weekly. The rationale for dose escalation of carfilzomib to 56mg/m2 is based on two findings: a) the 20/56mg/m2 dose escalation was well tolerated in the PX-171-007 trial and b) no dose limiting toxicities were seen with carfilzomib 20/27mg/m2 when combined with lenalidomide and dexamethasone in patients with RRMM who were heavily pre-treated, in the PX-171-006 and PX-171-009 trial. The rationale for assigning an equal number of patients between the ALLG sites and AMN sites is to avoid bias with respect to potential biological differences between patients in Asia and Australia/New Zealand.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients, ≥18 years of age
2. Relapsed and/or refractory multiple myeloma at study entry.
3. Patients must have evaluable multiple myeloma with at least one of the following (assessed within 21 days prior to registration):

   1. Serum M-protein ≥ 5 g/L, or
   2. Urine M-protein ≥ 200 mg/24 hour, or In patients without detectable serum or urine M-protein, serum free light chain (SFLC) > 100 mg/L (involved light chain) and an abnormal serum k/l ratio or For IgA patients whose disease can only be reliably measured by serum quantitative immunoglobulin (qIgA) ≥ 7500 mg/L (7.5 g/L).
4. Received one, but no more than three prior treatment regimens or lines of therapy for multiple myeloma. (Induction therapy followed by stem cell transplant and consolidation/maintenance therapy will be considered as one line of therapy).
5. Eastern Cooperative Oncology Group (ECOG) Performance Status 0-2.
6. Adequate hepatic function within 28 days prior to registration with bilirubin < 1.5 times the upper limit of normal (ULN), and aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 3 times the ULN.
7. LVEF ≥ 40%.
8. Absolute neutrophil count (ANC) ≥ 1000/mm3 (or 1000 cells/L) within 21 days prior to registration. Screening ANC should be independent of growth factor support for ≥ 1 week.
9. Platelet count ≥ 50,000 cells/mm3 (≥ 30,000 cells/mm3 if myeloma involvement in the bone marrow is > 50%) within 21 days prior to registration. Patients should not have received platelet transfusions for at least 1 week prior to obtaining the screening platelet count.
10. Calculated or measured creatinine clearance (CrCl) of ≥ 15 mL/min within 21 days prior to registration. Calculation should be based on the Cockcroft and Gault formula (Appendix 3)
11. Written informed consent in accordance with federal, local, and institutional guidelines.
12. Female patients of child-bearing potential (FCBP) must have negative serum pregnancy test within 21 days prior to registration and agree to use an effective method of contraception during and for 3 months following last dose of drug.
13. Male patients must use an effective barrier method of contraception during study and for 3 months following the last dose if sexually active with a FCBP.

Exclusion Criteria:

1. Chemotherapy with approved or investigational anticancer therapeutics within 21 days prior to registration, with the exception of dexamethasone up to 160mg or equivalent every 4 weeks.
2. Previous treatment with carfilzomib.
3. Focal radiation therapy within 7 days prior to registration. Radiation therapy to an extended field involving a significant volume of bone marrow within 21 days prior to registration (i.e., prior radiation must have been to less than 30% of the bone marrow).
4. Active congestive heart failure (New York Heart Association [NYHA] Class III to IV), symptomatic ischemia, or conduction abnormalities uncontrolled by conventional intervention. Myocardial infarction within four months prior to registration.
5. Acute active infection requiring systemic antibiotics, antiviral (except antiviral therapy directed at hepatitis B) or antifungal agents within 14 days prior to registration.
6. Known HIV seropositive and/or untreated hepatitis B (patients with hepatitis B surface antigen [HBsAg] and core antibody [HBcAb] are eligible if receiving adequate antiviral therapy directed at hepatitis B).
7. Patients with known cirrhosis.
8. Active malignancy, that is expected to require treatment with chemotherapy within one year, or results in a life expectancy less than one year.
9. Female patients who are pregnant or lactating.
10. Known history of allergy to Captisol (a cyclodextrin derivative used to solubilize carfilzomib)
11. Patients with hypersensitivity to carfilzomib, velcade, boron, or mannitol.
12. Patients with pleural effusions requiring thoracentesis or ascites requiring paracentesis within 14 days prior to registration.
13. Significant neuropathy (Grades 3-4, or Grade 2 with pain) within 14 days prior to registration.
14. Any other clinically significant medical disease or psychiatric condition that, in the Investigator's opinion, may interfere with protocol adherence or a patient's ability to give informed consent.

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-09-13 (Actual); Primary Completion 2019-06-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | 5 years or until disease progression
  To assess the progression free survival (PFS) in patients with RRMM who have had 1 to 3 prior lines of therapies, treated with combination carfilzomib, thalidomide and dexamethasone (CaTD)

SECONDARY OUTCOMES:
Overall survival (OS) | 5 years
  Defined as the duration from the start of treatment (C1D1) to death from any cause.
Overall Rate of Response (ORR) | anytime from commencement of treatment to the end of study baseline until disease progression, unmanageable adverse event or death, whichever occurs first, approximately up to 3 years
  percentage of patients enrolled that achieve a complete response (CR), or stringent complete response (sCR), or very good partial response (VGPR), or partial response (PR) based on the International Myeloma Working Group criteria
Duration of response (DOR) | 5 years
  Defined as the duration from the first response to the time of progression. Duration of response will be censored by deaths due to causes other than progression
Time to progression (TTP) | 5 years
  Defined as the duration from the start of treatment (C1D1) to disease progression or relapse based upon IMWG criteria, with deaths due to causes other than progression censored
Number of Participants affected by Adverse Events | Baseline up to 4 Weeks after the last dose of study drug administration
  An AE is any untoward medical occurrence attributed to study drug in a participant who received study drug. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Quality of life of participants on treatment | Approximately 3 years
  Health-related quality of life (HR-QOL) will be measured by the European standardized instrument EuroQoL EQ-5D-5L

CONTACTS AND LOCATIONS:
Overall Officials: Wee Joo Chng, Principal Investigator — National University Hospital, Singapore
Locations (4):
- Queen Mary Hospital, Hong Kong, Hong Kong
- National University Hospital, Singapore, Singapore
- South Korea, South Korea
- National Taiwan University, Taipei, Taiwan

REFERENCES:
- [Derived] Ninkovic S, Harrison SJ, Lee JJ, Murphy N, Lee JH, Estell J, Chen VM, Horvath N, Kim K, Eek R, Augustson B, Bang SM, Huang SY, Rajagopal R, Szabo F, Engeler D, Butcher BE, Mollee P, Durie B, Chng WJ, Quach H. Carfilzomib, thalidomide, and dexamethasone are safe and effective in relapsed and/or refractory multiple myeloma: final report of the single-arm, multicenter, phase II ALLG MM018/AMN002 study. Haematologica. 2024 Jul 1;109(7):2229-2238. doi: 10.3324/haematol.2023.284238. PMID 38235519